CLINICAL TRIAL: NCT03903081
Title: A Phase I, Single Center, Randomized, Double-blind, Placebo-controlled, Single & Multiple Ascending Dose Study to Access the Tolerability and Pharmacokinetics of HEC110114 Tablets in Healthy Adult Subjects
Brief Title: The Tolerability and Pharmacokinetics Study of HEC110114 Tablets in Healthy Adult Subjects
Acronym: HEC110114
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HEC110114-P-01
Record Dates: First submitted 2019-04-03; First posted 2019-04-04 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2019-04

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- 100 mg single dose (Experimental): It includes two groups, one group is pilot study, healthy subjects receive a single dose of 100 mg HEC110114 tablet (N=2) . Another group is formal study, healthy subjects receive a single dose of 100 mg HEC110114 tablet (N=8) or matching placebo (N=2)
  Interventions: Drug: HEC110114 tablet; Drug: Placebo Oral Tablet
- 300 mg single dose (Experimental): Healthy subjects, receiving a single dose of 300 mg HEC110114 tablet (N=8) or matching placebo (N=2)
  Interventions: Drug: HEC110114 tablet; Drug: Placebo Oral Tablet
- 600 mg single dose (Experimental): Healthy subjects, receiving a single dose of 600 mg HEC110114 tablet (N=8) or matching placebo (N=2)
  Interventions: Drug: HEC110114 tablet; Drug: Placebo Oral Tablet
- 800 mg single dose (Experimental): Healthy subjects, receiving a single dose of 800 mg HEC110114 tablet (N=16) or matching placebo (N=2) under fed or fasted conditions, this group is a two-sequence, two-period crossover study
  Interventions: Drug: HEC110114 tablet; Drug: Placebo Oral Tablet
- 1000 mg single dose (Experimental): Healthy subjects, receiving a single dose of 1000 mg HEC110114 tablet (N=8) or matching placebo (N=2)
  Interventions: Drug: HEC110114 tablet; Drug: Placebo Oral Tablet
- 1200 mg single dose (Experimental): Healthy subjects, receiving a single dose of 1200 mg HEC110114 tablet (N=8) or matching placebo (N=2)
  Interventions: Drug: HEC110114 tablet; Drug: Placebo Oral Tablet
- 1600 mg single dose (Experimental): Healthy subjects, receiving a single dose of 1600 mg HEC110114 tablet (N=8) or matching placebo (N=2)
  Interventions: Drug: HEC110114 tablet; Drug: Placebo Oral Tablet
- 600 mg multiple doses (Experimental): Healthy subjects, receiving 600 mg HEC110114 tablet (N=10) or placebo(N=2) once daily (q.d.) for 7 days
  Interventions: Drug: HEC110114 tablet; Drug: Placebo Oral Tablet
- 800 mg multiple doses (Experimental): Healthy subjects, receiving 800 mg HEC110114 tablet (N=10) or placebo(N=2) once daily (q.d.) for 7 days
  Interventions: Drug: HEC110114 tablet; Drug: Placebo Oral Tablet
- 1000 mg multiple doses (Experimental): Healthy subjects, receiving 1000 mg HEC110114 tablet (N=10) or placebo(N=2) once daily (q.d.) for 7 days
  Interventions: Drug: HEC110114 tablet; Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: HEC110114 tablet — administered orally once daily
Drug: Placebo Oral Tablet — Placebo will be administered orally at a dose and frequency matched to HEC110114

SUMMARY:
A Phase I, Single Center, Randomized, Double-blind, Placebo-controlled, Single & Multiple Ascending Dose Study to Access the Tolerability and Pharmacokinetics of HEC110114 Tablets in Healthy Adult Subjects

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent form before the trial and fully understand the contents of the trial, the process and possible adverse reactions
* Be able to complete the study according to the trail protocol
* Subjects (including partners) have no pregnancy plan within six months after the last dose of study drug and voluntarily take effective contraceptive measures
* Male subjects and must be 18 to 45 years of age inclusive
* Body weight ≥ 50 kg and body mass index（BMI）between 18 and 28 kg/m2, inclusive
* Physical examination and vital signs without clinically significant abnormalities.

Exclusion Criteria:

* Use of >5 cigarettes per day during the past 3 months
* Allergies constitution ( multiple drug and food allergies)
* History of alcohol abuse (14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of spirits or 100 mL of wine)
* Donation or loss of blood over 450 mL within 3 months prior to screening
* 12-lead ECG with clinically significant
* Positive for Viral hepatitis (including hepatitis B and C), HIV and syphilis
* Subjects deemed unsuitable by the investigator for any other reason.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2019-10-29 (Actual); Study Completion 2019-10-29 (Actual)

PRIMARY OUTCOMES:
Adverse Events | From Days 1-12
  Percentage of Participants with Adverse Events

SECONDARY OUTCOMES:
Cmax | At pre-defined intervals from Days 1-12
  Maximum Observed Plasma Concentration
Tmax | At pre-defined intervals from Days 1-12
  Time to Maximum Observed Plasma Concentration
AUClast | At pre-defined intervals from Days 1-12
  Area Under the Plasma Concentration vs Time Curve to Last Measurable Concentration
AUC0-∞ | At pre-defined intervals from Days 1-12
  Area Under the Plasma Concentration vs Time Curve Extrapolated to Infinity
T1/2 | At pre-defined intervals from Days 1-12
  Apparent Half-Life
CL/F | At pre-defined intervals from Days 1-12
  Clearance (CL/F) of HEC110114
Cmin | At pre-defined intervals from Days 1-11 for MAD
  Trough Plasma Concentration of HEC110114

CONTACTS AND LOCATIONS:
Overall Officials: Yanhua Ding, Doctor, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China